CLINICAL TRIAL: NCT00385047
Title: Phase I/IIa Study of the Safety, Immunogenicity and Preliminary Efficacy After Sporozoite Challenge of FMP2.1/AS01B and FMP2.1/AS02A Candidate Malaria Vaccines Administered Intramuscularly at Months 0, 1, and 2 in Malaria-naive Adults Living in the United States
Brief Title: A Study to Determine Whether 2 Investigational Malaria Vaccines Are Safe, Protective Against Malaria in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); GlaxoSmithKline (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR 1280; A-13949 (Other: WRAIR Protocol ID); ETrack Protocol No. 104936 (Other: E-Track); MAL-045 (Other: GSK); #20060900 (Other: Internal)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Malaria
Keywords: malaria; vaccine; AMA-1 (apical membrane antigen-1); efficacy
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): FMP 2.1 50 μg FMP2.1/AS01B
  Interventions: Biological: Group A FMP2.1/AS01B
- Group B (Experimental): FMP 2.1 50 μg FMP2.1/AS02A
  Interventions: Biological: Group B FMP2.1/AS02A

INTERVENTIONS:
Biological: Group A FMP2.1/AS01B
  Other Names: FMP 2.1 50 μg FMP2.1/AS01B
  Arms: Group A
Biological: Group B FMP2.1/AS02A
  Other Names: FMP 2.1 50 μg FMP2.1/AS02A
  Arms: Group B

SUMMARY:
The purpose of this study is to determine whether 2 investigational malaria vaccines are safe as well as protective against malaria in adults living in the United States

DETAILED DESCRIPTION:
35 volunteers aged 18 to 50 years will be enrolled to receive one of 2 investigational malaria vaccines. The vaccines are made of a malaria protein FMP2.1 mixed in 2 different adjuvants (AS01B and AS02A). Five volunteers will get a small (10 µg) dose of FMP2.1/AS01B since this vaccine has not yet been in humans. If it is safe, then 15 volunteers will get 50 µg FMP2.1 in AS02A and 15 will get 50 µg FMP2.1 in AS01B. All vaccines are given IM in the deltoid of the non-dominant arm, every 1 month for 3 months. After vaccination, the subjects will follow up at clinical trials for evaluation of any adverse events.

20 vaccinees (10 from each 50 µg vaccine group) will undergo primary sporozoite challenge 14-30 days after dose 3 via bite of 5 malaria-infected mosquitoes. All subjects will have a blood slide prepared and read to check for asexual P. falciparum parasitemia at least once daily beginning day 5 post challenge. Beginning on day 10 post challenge, subjects will check into a designated hotel, where 24 hour evaluation and care will be available for 10 nights. After this hotel phase, there will be follow-up visits to ensure there are no late developments of malaria in those who have not fallen ill (and thus are considered protected).

Any subject who tests positive for malaria will be treated with chloroquine. Efficacy readouts are complete protection or significant delay in patency defined as >2 days than the median prepatent period for the 6 infectivity controls. These 6 controls receive no vaccine and are enrolled for malaria-challenge only in order to provide comparison group for vaccinated individuals.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant female 18 to 50 years of age (inclusive) at the time of screening
* Written informed consent obtained from the participant before screening procedures
* Free of clinically significant health problems as established by medical history and clinical examination before entering into the study*
* Available to participate for duration of study (approximately five months, not including screening)
* If the participant is female, she must be of non-childbearing potential, i.e., either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or Depo-Provera®) during this study, have a negative pregnancy test at the time of each immunization, and must agree to continue such precautions for two months after completion of the immunization series and the malaria challenge.
* Prior to entry into this study, participants must score at least 80% correct on a short multiple-choice quiz that assesses their understanding of this study. If they do not score 80% on the initial quiz, the protocol information will be reviewed with them to ensure comprehension and they will have the opportunity to retest. Participants who fail the Comprehension Assessment for the second time will not be enrolled.

Exclusion Criteria:

* Prior receipt of an investigational malaria vaccine
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization or planned use during the study period, or receipt of investigational vaccine containing 3-D MPL and/or QS-21 at any time in the past (Have you received an experimental vaccine with a GSK adjuvant in the past?)
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of immunization. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Chronic use of antibiotics with anti-malarial effects (e.g., tetracyclines for dermatologic patients, sulfa for recurrent urinary tract infections, etc.)
* Planned administration of a vaccine not foreseen by the study protocol 30 days prior to or after the first immunization
* History of malaria chemoprophylaxis within 60 days prior to immunization
* Any history of malaria
* Known exposure to malaria within the previous 12 months
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* History of allergic disease or reactions to any vaccine
* Chronic or active neurologic disorders including seizures, excluding a single febrile seizure as a child
* History of splenectomy
* Acute disease at the time of enrollment (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., oral temperature < 37.5°C/99.5°F).
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Personal medical histories including the following diagnoses: systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, scleroderma, vasculitis, and multiple sclerosis
* Seropositive for hepatitis B surface antigen or hepatitis C antibody
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Elevated serum creatinine, defined in this study as greater than or equal to 1.7 mg/dL in males and 1.4 mg/dL in females
* Significant unexplained anemia: hematocrit < 35%
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period
* Pregnant or lactating female or female who intends to become pregnant during the study
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV (Diagnostic and Statistical Manual of Mental Disorders- 4th edition)
* Chronic or active illicit and/or intravenous drug use
* History of severe anaphylactic reactions to mosquito bites
* History of psoriasis (given its interaction with chloroquine)
* Any history of anaphylaxis in reaction to immunization
* History of allergy to nickel, imidazole or tetracycline group of antibiotics
* History of sickle cell disease or sickle cell trait
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 1 year

SECONDARY OUTCOMES:
Anti-AMA-1 antibody titers during Immunization Phase | Up to 70 days
Anti-AMA-I antibody titers during Challenge Phase | Up to 90 days
Anti-AMA-I antibodies as percent parasite growth inhibition during Immunization Phase | Up to 70 days
Anti-AMA-I antibodies as percent parasite growth inhibition during Challenge Phase | Up to 90 days
Time to parasitemia development after primary challenge following administration of the FMP2.l/ASOIB and FMP2.l /AS02A | Up to 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Michele D. Spring, MD, M.S.P.H., Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Clinical Trials Center, Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Background] Dutta S, Lalitha PV, Ware LA, Barbosa A, Moch JK, Vassell MA, Fileta BB, Kitov S, Kolodny N, Heppner DG, Haynes JD, Lanar DE. Purification, characterization, and immunogenicity of the refolded ectodomain of the Plasmodium falciparum apical membrane antigen 1 expressed in Escherichia coli. Infect Immun. 2002 Jun;70(6):3101-10. doi: 10.1128/IAI.70.6.3101-3110.2002. PMID 12011004
- [Derived] Spring MD, Cummings JF, Ockenhouse CF, Dutta S, Reidler R, Angov E, Bergmann-Leitner E, Stewart VA, Bittner S, Juompan L, Kortepeter MG, Nielsen R, Krzych U, Tierney E, Ware LA, Dowler M, Hermsen CC, Sauerwein RW, de Vlas SJ, Ofori-Anyinam O, Lanar DE, Williams JL, Kester KE, Tucker K, Shi M, Malkin E, Long C, Diggs CL, Soisson L, Dubois MC, Ballou WR, Cohen J, Heppner DG Jr. Phase 1/2a study of the malaria vaccine candidate apical membrane antigen-1 (AMA-1) administered in adjuvant system AS01B or AS02A. PLoS One. 2009;4(4):e5254. doi: 10.1371/journal.pone.0005254. Epub 2009 Apr 23. PMID 19390585